CLINICAL TRIAL: NCT03663179
Title: A Pilot Study of Repetitive Transcranial Magnetic Stimulation for Adult ADHD
Brief Title: Transcranial Magnetic Stimulation for Attention Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 826586
Record Dates: First submitted 2018-08-02; First posted 2018-09-10 (Actual); Results first posted 2019-10-28 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Attention Deficit Disorder With Hyperactivity (ADHD)
Keywords: ADHD; TMS
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active TMS (Experimental): Participants will receive 20 sessions of active TMS targeting the left DLPFC.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- Sham TMS (Sham Comparator): Participants will receive 20 sessions of sham TMS over the left DLPFC.
  Interventions: Device: Sham Transcranial Magnetic Stimulation (Sham TMS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — A MagPro R30 (Magventure, Inc., Copenhagen, Denmark) device with a Cool-B65 A/P figure 8 coil will be used to deliver TMS. This coil has an active side and a sham side, and can be used to perform double-blinded studies. TMS will be administered at 10 Hertz (Hz) with an intensity of 120% of patient resting motor threshold. Stimulation will be delivered to the left dorsolateral prefrontal cortex using 20 sec cycles (i.e., 5 sec train with 15 sec inter train interval). Subjects will receive 80 trains per session for a total of 4000 pulses per session (~26 min sessions). Twenty sessions will be completed on sequential weekdays (5 days per week for 4 weeks).
  Arms: Active TMS
Device: Sham Transcranial Magnetic Stimulation (Sham TMS) — A MagPro R30 (Magventure, Inc., Copenhagen, Denmark) device with a Cool-B65 A/P figure 8 coil will be used to deliver TMS. This coil has an active side and a sham side, and can be used to perform double-blinded studies. For sham stimulation, the sham side of the coil is positioned toward the participant's scalp. The sham coil is designed to mimic the appearance and sound of active TMS stimulation, but is equipped with a magnetic shield that reduces the strength of the field by approximately 80%. This reduction in field strength ensures that no neural stimulation occurs. Twenty sessions will be completed on sequential weekdays (5 days per week for 4 weeks).
  Arms: Sham TMS

SUMMARY:
This study will test the effects of transcranial magnetic stimulation (TMS) on clinical measures of ADHD symptoms.

DETAILED DESCRIPTION:
Attention Deficit Hyperactivity Disorder (ADHD) is characterized by symptoms of impulsivity, inattention, and hyperactivity that emerge in childhood and frequently persist into adulthood. These symptoms are accompanied by deficits in cognitive control and risky decision making that can lead to negative psychosocial and health-related outcomes. With advances in the neuroimaging field, researchers are learning where and how self-control over decisions and behaviors is executed in the brain. This work points to the central role of neural activity in the dorsolateral prefrontal cortices (DLPFC) in self-control processes that contribute to healthy choices. Emerging evidence shows that activity in the prefrontal cortices and cognitive control circuits can be modulated using a noninvasive and safe intervention: repetitive TMS. This within-subject proof of concept study will investigate whether 20 sessions of TMS (versus sham stimulation) can enhance executive cognitive function in adults with ADHD.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants will be:

1. Healthy males and females who are between 18 and 65 years of age with an ADHD diagnosis (meet diagnostic criteria for ADHD on the SCID-5 module for adult ADHD).
2. Planning to live in the area for at least the next 6 weeks;
3. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent and HIPAA form;
4. Able to communicate fluently in English (speaking, writing, and reading).

Exclusion Criteria:

Subjects who present and/or self-report with the following criteria at any point during study participation will not be eligible to participate in the study:

Alcohol/Drugs:

1. History or current diagnosis or treatment for alcohol or drug abuse (as reported during phone screen);
2. Positive breath alcohol concentration test (BrAC greater than or equal to 0.01) at intake;
3. A positive urine drug screen for cocaine, phencyclidine (PCP), amphetamines, methamphetamines, benzodiazepines, methadone, and/or barbiturates at Intake, Baseline, or Sessions 5, 10, 15 or 20.

Medication:

Current use or recent discontinuation (within the past 6 months at the time of Intake) of:

1. Gamma-Aminobutyric Acid (GABA)-ergic medications
2. Glutamatergic medications
3. Any medication for the treatment of ADHD
4. Benzodiazepines
5. Any medication that is known to lower the seizure threshold (e.g.,clozapine, bupropion, tramadol, carbapenems, stimulants)
6. Any medication that could compromise participant safety as determined by the Principal Investigator and/or Study Physician

   Current use or recent discontinuation (within the last 14 days at the time of Intake) of:
7. Anti-psychotic medications
8. Nicotine replacement therapy (NRT)

   Daily use of:
9. Opiate-containing medications for chronic pain

Medical/Neuropsychiatric:

1. Women who are pregnant, planning a pregnancy, and/or breast feeding.
2. History of seizures, epilepsy, or history of epilepsy in first-degree relative
3. History of stroke or transient ischemic attack (warning stroke)
4. History of traumatic brain injury or self-report of brain or spinal tumor
5. History of head injury with unconsciousness lasting more than 5 minutes
6. Previous brain surgery
7. Any additional neurological condition that would likely reduce the safety of study participation, including central nervous system (CNS) vasculitis, intracranial tumor, intracranial aneurysm, multiple sclerosis or arteriovenous malformations
8. History of tinnitus
9. History of diabetes mellitus
10. History of atherosclerotic vascular disease
11. A medically unstable cardiopulmonary or metabolic disorder
12. Increased risk for myocardial infarction or other major cardiopulmonary complications.
13. Any uncorrected visual impairment or abnormality
14. Self-reported history, current diagnosis of psychosis or symptoms consistent with a mood disorder based upon the Structured Clinical Interview for DSM-5 (SCID); including schizophrenia, mania, bipolar disorder, an eating disorder, obsessive compulsive disorder, an anxiety disorder, major depression (subjects with a history of major depression but in remission for past 6 months are eligible).

TMS-related:

1. Subjects with ferromagnetic material in or in close proximity to the head (with the exception of oral dental devices)
2. Implanted devices (including vagus nerve stimulator (VNS), deep brain stimulator (DBS), pacemakers, spinal cord stimulators, medication pumps, ventriculo peritoneal shunts, defibrillators, intracardiac lines)
3. Self-report of any skull fracture or opening
4. A disturbance in normal sleep patterns/sleep deprivation

General Exclusion:

1. Any medical condition, illness, disorder, or concomitant medication that could compromise participant safety or treatment, or affect clinical or cognitive outcomes, as determined by the Principal Investigator
2. Inability to complete study tasks and provide quality data, as determined by the Principal Investigator
3. Low or borderline intellectual functioning - determined by a score of less than 90 on the Shipley Institute of Living Scale (SILS) (administered at Intake Visit). The SILS correlates with the Wechsler Adult Intelligence Scale-Revised (WAIS-R) Estimated Intelligence Quotient (IQ) Test
4. Inability to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2020-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Loughead, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active TMS | Sham TMS
Started | 18 | 14
Completed | 14 | 13
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Revealed exclusionary condition | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active TMS | Sham TMS | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (9.9) | 36.0 (6.0) | 34.4 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 9 | 9 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 10 | 9 | 19
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Education [Count of Participants; unit: Participants]
  high school/some college | 7 | 4 | 11
  college graduate | 7 | 9 | 16
Smoking Status [Count of Participants; unit: Participants]
  smokers | 4 | 2 | 6
  non-smokers | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Performance on Conners Adult ADHD Rating Scale - Self-Report: Long Version (ADHD Symptoms)
Description: ADHD symptoms will be assessed using the well-validated Conners Adult ADHD Rating Scale - Self-Report: Long Version (CAARS-S:L). The CAARS-S:L is a 66-item rating scale designed to assess ADHD symptoms in adults. The scale contains multiple subscales to assess Diagnostic and Statistical Manual of Mental Disorders 4th edition (DSM-IV) specified ADHD criteria as well as other facets of ADHD such as inattention/memory problems, hyperactivity/restlessness, impulsivity/emotionality, and problems with self-concept. Subscale results are converted to T-scores (range: 25-90), where 50 is the standardized population mean and every 10 points indicates one standard deviation from the mean. Higher values generally indicate more difficulties with ADHD symptoms. This measure will be administered at baseline at at the end of 4 weeks of treatment. The primary outcome will be the change from baseline to week 4.
Time Frame: Baseline and week 4
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Active TMS | Sham TMS
Number analyzed (Participants) | 14 | 13
t-score | -4.4 (9.4) | -5.1 (7.6)

2. Secondary Outcome: Change in Performance on Conners Continuous Performance Task (Sustained Attention)
Description: The Conners Continuous Performance Task (Conners CPT) will be administered and baseline and weekly during the treatment period to assess sustained attention. In this task, participants are shown a series of letters on a computer screen and are asked to press the spacebar in response to all letters except for the letter X. The primary outcome for the Conners CPT is the change in number of commission errors (e.g., false positives) from baseline to week 4.
Time Frame: Baseline and week 4
Measure: Mean (Standard Deviation); unit: Commission Errors
Arm/Group | Active TMS | Sham TMS
Number analyzed (Participants) | 14 | 13
Commission Errors | -16.2 (17.6) | -4.8 (18.0)

ADVERSE EVENTS:
Time Frame: Baseline until end of treatment, an average of 4 weeks.
Arm/Group | Active TMS | Sham TMS
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/14
Other Adverse Events (participants affected / at risk) | 4/18 | 1/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TMS (N=18) | Sham TMS (N=14)
Sleep disturbance (General disorders) | 1 (1) | 0 (0) — Participant experienced insomnia several times during the first week of treatment and revealed a history of insomnia prior to enrollment.
allergic reaction (Immune system disorders) | 1 (1) | 0 (0) — Participant unknowingly consumed peanuts while at their personal gym and experienced an allergic reaction.
Visual disturbance (Eye disorders) | 0 (0) | 1 (1) — Participant reported seeing a white flash while completing computer tasks after receiving her 10th session of TMS.
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Participant diagnosed with tendinitis in left foot and needed to wear a boot.
Depression symptoms (Psychiatric disorders) | 1 (1) | 0 (0) — Participant reported depression symptoms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-29): https://cdn.clinicaltrials.gov/large-docs/79/NCT03663179/Prot_SAP_000.pdf